CLINICAL TRIAL: NCT04493957
Title: Evaluation of a Psycho-educational Program Based on the Prevention of the Risks Related to the Impact of Cognitive Disorders on Driving in Geriatrics and Neurology
Brief Title: Evaluation of an Educational Program in the Prevention of the Driving Risks in Patients With Neurocognitive Disorders : ACCOMPAGNE
Acronym: ACCOMPAGNE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: new law making inclusion impossible
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 69HCL19_0676
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Driving Habits Patients; Cognitive Impairment
Keywords: driving habits; cognitive impairment; prevention; educational intervention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- educational intervention (Experimental): Patients and caregivers included in the "ACCOMPAGNE Education Program" group will benefit from seven group workshops spread over three half-days (once a week over 3 consecutive weeks), animated in pairs, each lasting approximately one and a half hours. and using educational pedagogical methods.
  Interventions: Behavioral: ACCOMPAGNE Education Program
- Control group (Active Comparator): Patients and caregivers included in the "Control" group will receive the usual recommendations for driving, issued by their referring doctor in memory consultation during the diagnostic announcement process or during the follow-up of their illness.
  Interventions: Behavioral: Usuals recommandations

INTERVENTIONS:
Behavioral: ACCOMPAGNE Education Program — The following workshops will be organised :
  * Presentation workshop
  * Cognitive skills" workshop
  * Perception and Environment workshop
  * Responsibilities workshop
  * Representation workshop -
  * Caregivers workshop,
  * Solutions workshop
  Arms: educational intervention
Behavioral: Usuals recommandations — Recommendations consist of a description of the cognitive and sensorimotor risk factors specific to the patient for driving and advice for the adaptation of driving or the recommendation of the stopping of driving. It is usually served by oral or written to the patient, with mention in the patient's file of the recommendation and issued in the presence of his close companion.
  Arms: Control group

SUMMARY:
ACCOMPAGNE study proposes to evaluate an educational program for the patient / caregiver dyad, intended to accompany the patient towards the implementation of self-regulation strategies in the driving activity. The program, based on group workshops with the presence of the patient and the caregiver, is led by an interdisciplinary team. It follows all the intervention recommendations described in the literature: to make the patient a decision-maker, to allow advanced planning of discussions between the family member and the caregiver, to give information on the consequences of TNCs and sensory disorders. This program provides psychological support in the management of the problems and the mourning of a future cessation of the driving activity, an awareness of the risky and avoidable situations, information on alternative solutions and available resources in the event of reduced driving. The program is created to support the implementation of self-regulation strategies for safe driving and a gradual reduction of driving activity. This study may be included in Measure 5 of the Neuro-Degenerative Diseases Plan (PMND) 2014-2019. This plan recommends to strengthen the self-management of patients and their relatives in the disease.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50 and 95 years-old
* hold a driving license,
* drive at least twice a week,
* to have given free and informed consent,
* present a diagnosis of major or minor CNS according to DSM V, whose clinically probable or definite etiology is Alzheimer's or related or vascular disease,
* have a result in the Mini Mental State Examination (MMSE) greater than 18,
* have the ability to speak orally enough or write enough to perform clinical evaluations and workshops, be accompanied by a family member present at least 4 hours a week.

Criteria for inclusion of carers:

* to be a caregiver helping the patient for activities of daily living,
* to have given their free and informed consent,
* have the ability to speak orally and write enough to perform clinical assessments.

Exclusion Criteria:

* have a major psychiatric history, history of alcoholism, anti-depressant
* have sensory problems preventing participation in workshops,
* be affected by any debilitating pathology compromising the health of the patient in the short and medium term,
* be unable to express consent. Criteria for non-inclusion of caregivers: have sensory disturbances preventing participation in workshops.

Recruited patients and caregivers should have been informed and signed a consent.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
short term setting up self-regulation strategies | at 2 months
  The score on the Driver Perception and Practices Questionnaires : DPPQ's "Current Self Regulatory Practices" subscale completed by the patient will be the primary outcome. The scores will be compared at 2 months between the control group and the experimental group. The Current Self Regulatory Practices subscale consists of 8 questions about how often participants set up self-regulation strategies (wait for the rain to stop before driving, ask someone to travel with them rather than drive alone, look for parking to avoid niches, avoid turning left in traffic, avoid taking the freeway, avoid driving at rush hour, avoid driving in crowded places, avoid driving the night). A four-point scale (0: never, 1: rarely, 2: sometimes, 3: often) collects the frequency. The score is calculated by summing the response values on the eight driving situations creating a total score ranging from 0 (never execute any of these strategies) to 24 (often performs all strategies).

SECONDARY OUTCOMES:
long term setting up self-regulation strategies | six months
  The score on the Driver Perception and Practices Questionnaires : DPPQ's "Current Self Regulatory Practices" subscale. The scores will be compared to 6 months between the control group and the experimental group. A four-point scale (0: never, 1: rarely, 2: sometimes, 3: often) collects the frequency.
Indicators of driving changes | two months and six months
  a composite score with the first part of the Driving Habits Questionnaire (DHQ) used to collect driving habits (number of journeys per day / week / month, number of kilometers traveled, confidence in driving skills) and the other sub- DPPQ scales. The Driver Perception and Practices Questionnaires (DPPQ) have a four-point scale (0: never, 1: rarely, 2: sometimes, 3: often) collects the frequency. the DHQ questionnaire have four-point scale (0 : never, 1 : without any difficulty, 2 : with some difficulty, 3: with moderate difficulty, 4 : with a lot of difficulty) another questions should be answered by yes or no, to assess driving habits.
Indicators of changes perceived by the caregiver | two months and six months
  a composite score with the Driver Perception and Practices Questionnaires (DPPQ) scale supplemented by the caregiver from the observations made on the patient's driving and the first part of the DHQ scale supplemented by the caregiver from the observations made he patient's driving. The DPPQ have a four-point scale (0: never, 1: rarely, 2: sometimes, 3: often) collects the frequency. The Driving Habits Questionnaire (DHQ) have four-point scale (0 : never, 1 : without any difficulty, 2 : with some difficulty, 3: with moderate difficulty, 4 : with a lot of difficulty) another questions should be answered by yes or no, to assess driving habits.
Indicators of awareness of driving difficulties | two months and six months
  score obtained in the second part of the Driving Habits Questionnaire (DHQ) : Driving Habits Questionnaire scale and comparison with the scores obtained on the driving simulator. The Driving Habits Questionnaire (DHQ) have four-point scale (0 : never, 1 : without any difficulty, 2 : with some difficulty, 3: with moderate difficulty, 4 : with a lot of difficulty) another questions should be answered by yes or no, to assess driving habits.
Indicators of Mood Effects of Conduct Modifications on the patient | two months and six months
  The Geriatric Depression Scale Scale 15 items (GDS 15). This scale consists of 15 questions to be answered by yes or no. 0 being the minimum score, 15 being the maximum score. The Geriatric Depression Scale was designed to look for depressive symptoms in older depressive symptoms in elderly subjects.
Indicators of quality of life effect of Conduct Modifications on the patient | two months and six months
  Quality of Life Quality of Life Alzheimer Disease (QoL-AD) Scale. This scale uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks in order to evaluate the quality of life of patients.
Indicators of Mood Effects of Conduct Modifications on the caregivers | two months and six months
  The Geriatric Depression Scale Scale 15 items (GDS 15). This scale consists of 15 questions to be answered by yes or no. 0 being the minimum score, 15 being the maximum score. The Geriatric Depression Scale was designed to look for depressive symptoms in older depressive symptoms in elderly subjects.
Indicators of quality of life effect of Conduct Modifications on the caregivers | two months and six months
  Quality of Life Quality of Life Alzheimer Disease (QoL-AD) Scale. This scale uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks in order to evaluate the quality of life of patients.
Indicators of burden caregiver effect of Conduct Modifications | two months and six months
  The Zarit scale.This scale uses a scale of 1-5 (never, rarely, sometimes, quite often or almost often) to assess hardship or burden assessment.
Indicators on the overall usefulness of the program | two months and six months
  The general utility of the program will be measured by adapting a questionnaire from Levasseur et al. (2014) study. This questionnaire focuses on several dimensions. The question is whether the participants found an interest in the program, whether the program allowed them to be more open to the issue of conduct and the link with cognitive disorders, and whether they acquired knowledge in this field. It is also important to know whether participants and caregivers are aware of post-program changes and the implementation of compensatory strategies. The questionnaire will also collect on a scale of Lickert the intention to stop driving at the moment (1: no intention to 4: important intention) as well as the driving cessation by the question "Have you stopped driving, if so, how long? ".
Indicators of program acceptability | two months
  Acceptability will be measured by analyzing the proportion of refusals to participate in the study, and enrollment at 2 months in the experimental group. The reason for refusals and stops during the educational sessions will be collected and analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Charpennes Hospital, Villeurbanne, France

REFERENCES:
- [Derived] Delphin-Combe F, Coste MH, Bachelet R, Llorens M, Gentil C, Giroux M, Paire-Ficout L, Ranchet M, Krolak-Salmon P. An innovative therapeutic educational program to support older drivers with cognitive disorders: Description of a randomized controlled trial study protocol. Front Neurol. 2022 Jul 18;13:901100. doi: 10.3389/fneur.2022.901100. eCollection 2022. PMID 35923824